CLINICAL TRIAL: NCT01737320
Title: Duration of Antibiotics for the Treatment of Gram-negative Bacilli Bacteremia - a Randomized Controlled Trial
Brief Title: Duration of Antibiotics for the Treatment of Gram-negative Bacilli Bacteremia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, dafna yahav, MD, a specialist in internal medicine and a specialist in the infectious disease unit, Principal investigator., Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0258-12-RMC
Record Dates: First submitted 2012-11-14; First posted 2012-11-29 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Gram Negative Bacteremia
Keywords: gram negative bacteremia; Duration of antibiotic treatment; safety; efficacy; short-course

ARMS (2):
- short-course (Experimental): antibiotic treatment stopped on day 7 if the patient has been afebrile for 48 hours and clinically stable. Continued hospitalization will be left to the discretion of the treating physician. Antibiotics will be restarted if fever recurs in at least 2 consecutive measurements above 38 or in cases of clinically or microbiologically documented infections.
  Interventions: Drug: short-course antibiotic treatment
- accepted prolonged antibiotic treatment (Active Comparator): antibiotic treatment continued for 14 days according to accepted hospital local guidelines. Duration of hospital stay will also be left to the discretion of the treating physician.
  Type of empiric antibiotic treatment and later, specific antibiotic treatment, will be chosen by the treating physicians in consultation with the infectious diseases unit.
  The decision on timing of switch to oral antibiotic therapy will also be left to the discretion of the treating physician.
  Interventions: Drug: accepted prolonged antibiotic treatment

INTERVENTIONS:
Drug: short-course antibiotic treatment — On day 7 of appropriate intravenous or oral antibiotic treatment for the bacteremic episode (day 1 is the first day of appropriate antibiotic therapy), patients will be randomized to:
  1. Intervention group - antibiotic treatment stopped on day 7
  2. Control group - antibiotic treatment continued for 14 days according to accepted hospital local guidelines.
  Arms: short-course
Drug: accepted prolonged antibiotic treatment
  Arms: accepted prolonged antibiotic treatment

SUMMARY:
The investigators plan an open label randomized controlled trial to compare short-course antibiotic therapy (<=7 days) versus longer treatment (>7 days). The investigators will include hospitalized patients with gram-negative bacteremia. The investigators primary objective is to investigate the safety and efficacy of short-course antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* patients with gram-negative aerobic bacilli bacteremia, defined as growth of a single gram-negative microorganism in one or more blood cultures, associated with evidence of infection (hyper- or hypothermia, a localized infection, sepsis or septic shock).
* We will include patients receiving appropriate antibiotic treatment for 7 days and are afebrile / not hypothermic for the last 48 hours. Both community and hospital acquired gram-negative bacteremias will be included, regardless of antibiotic susceptibility patterns. We will allow the inclusion of patients receiving less than 7 days if clinically stable and discharge from hospital is considered. We will then recruit the patient before discharge, if stable at least for 48 hours before randomization.

We will include the following sources of bacteremia:

1. Primary bacteremia / unknown source
2. Urinary tract
3. Abdominal
4. Respiratory tract
5. Central venous catheter(CVC), when the catheter was removed before randomization
6. Skin and soft tissue, including surgical site infection

Exclusion Criteria:

1. Gram-negative bacteremia due to specific infections as detailed here:

   1. Endocarditis / endovascular infections
   2. Necrotizing fasciitis
   3. Osteomyelitis
   4. Abdominal abscesses and other unresolved abdominal sources requiring surgical intervention (e.g., cholecystitis)
   5. Central nervous system infections
   6. Empyema
   7. CVC- related or CVC-associated bloodstream infections when the catheter is retained. We will permit the inclusion of patients with retained CVCs in whom the source of the bacteremia is not the CVC.
2. Polymicrobial growth in blood cultures involving gram-positive or anaerobes in addition to gram-negatives (defined as either growth of two or more different species of microorganisms in the same blood culture, or growth of different species in two or more separate blood cultures within the same episode (< 48 h) and with clinical or microbiological evidence of the same source).
3. Specific pathogens including:

   1. Salmonella spp.
   2. Brucella spp.
4. Immunosuppression, including:

   1. HIV infection
   2. Hematopoietic stem-cell transplantation
   3. Neutropenia on day of randomization or in the 48 hours prior to randomization. Patients with neutropenic fever at presentation that are afebrile and non-neutropenic in the 48 hours before randomization will be included.
5. Clinical instability during the 48 hours before randomization, defined as mean blood pressure<60 mmHg despite adequate fluid resuscitation or vasopressors support.
6. Repeated positive blood cultures for the same organism separated by at least 24 hours, regardless of antibiotic treatment. Patients with repeated isolates on the first 24 hours will be included.
7. Uncontrolled focus of infection: e.g. an abscess that was not drained sufficiently; non-drained moderate to severe hydronephrosis in a patient with bacteremia of urinary source; deep seated intra-abdominal infections that were not drained properly.
8. Fever > 38.0C measured at least twice in the 48 h prior to recruitment; or > 38.5C once during the 48 h; or hypothermia <35.5C measured once during the 48 h.
9. Previous enrollment in this trial
10. Concurrent participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 2013-01; Primary Completion 2018-03 (Actual); Study Completion 2018-03-04 (Actual)

PRIMARY OUTCOMES:
composite of the following | Until day 90 after randomization
  The primary outcome is a composite of the following outcome measures
All -cause mortality | Until day 90 after randomization
  All- cause mortality
Treatment Failure | Until day 90 after randomization
  Failure including any of the following:
  1. Relapse: a recurrent bacteraemia due to the same microorganism occurring from day of randomization and until day 9013
  2. Local suppurative complication that was not present at infection onset (e.g. renal abscess in pyelonephritis, empyema in pneumonia)
  3. Distant complications of initial infection, defined by growth of the same bacteria as in the initial bacteremia
Hospital re-admissions or extended hospitalization | Until day 90 after randomization
  We will define re-admission as a new hospitalization for any cause occurring more than14 days from start of appropriate antibiotic treatment. Patients hospitalized after day 14 (were never discharged or 7-day regimen who were readmitted between days 7-14) will be counted as failures for this outcome.
  We will define re-admission as a new hospitalization for any cause occurring more than14 days from start of appropriate antibiotic treatment. Patients hospitalized after day 14 (were never discharged or 7-day regimen who were readmitted between days 7-14) will be counted as failures for this outcome.

SECONDARY OUTCOMES:
Clostridium difficile associated diarrhea | Until day 30 after randomization
  Clostridium difficile associated diarrhea
Development of Antibiotic resistance | Until day 30 after randomization
  Development of resistance, defined as clinical isolates resistant to antibiotics previously used in the bacteremia episode. Surveillance sampling will not be conducted.
Carriage of carbapenem resistant Klebsiella pneumonia. | Until day 30 after randomization
  Carriage of carbapenem resistant Klebsiella pneumonia (screened routinely)
Total in hospital days | Until day 90 after randomization.
  Total in hospital days within 30 and 90 days
Total antibiotic days | Until day 30 after randomization
  Total antibiotic days
Adverse events | Until day 30 after randomization
  * Any diarrhea
  * Liver function test abnormalities, defined as elevated bilirubin x 1.5 of upper limit of normal or transaminases x 2.5 of upper limit of normal
  * Antibiotic rash
  * Acute kidney injury - defined according to RIFLE criteria as increased creatinine level x 1.5 from baseline or glomerular filtration rate (GFR) decrease >25% or urine output of <0.5 ml/kg/h for 6 hours22
Infection caused by other than gram-negative bacteremia | Until day 90 after randomization
  Development of either clinically or microbiologically documented infection other than gram-negative bacteremia. We will use the 2008 CDC/NHSN surveillance definitions of health-care associated infections for bacterial infections
Number of hospital re-admissions | Until day 90 after randomization
  Number of hospital re-admissions until day 90
Functional capacity and time to return to baseline activity | Until day 30 after randomization
  Functional capacity and time to return to baseline activity

CONTACTS AND LOCATIONS:
Overall Officials: Dafna Yahav, MD, Principal Investigator — Rabin Medical Center
Locations (3):
- Israel (2):
  - Rambam Health Care Center, Haifa
  - Rabin medical center, Beilinson Hospital, Petah Tikvah
- Policlinico di Modena, Italy, Modena, Emilia-Romagna, Italy

REFERENCES:
- [Derived] Yahav D, Franceschini E, Koppel F, Turjeman A, Babich T, Bitterman R, Neuberger A, Ghanem-Zoubi N, Santoro A, Eliakim-Raz N, Pertzov B, Steinmetz T, Stern A, Dickstein Y, Maroun E, Zayyad H, Bishara J, Alon D, Edel Y, Goldberg E, Venturelli C, Mussini C, Leibovici L, Paul M; Bacteremia Duration Study Group. Seven Versus 14 Days of Antibiotic Therapy for Uncomplicated Gram-negative Bacteremia: A Noninferiority Randomized Controlled Trial. Clin Infect Dis. 2019 Sep 13;69(7):1091-1098. doi: 10.1093/cid/ciy1054. PMID 30535100